CLINICAL TRIAL: NCT00187798
Title: Impact of Genetics on Metformin Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 928
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: Healthy Control Twins
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Other): Metformin HCl
  Interventions: Drug: Metformin HCl

INTERVENTIONS:
Drug: Metformin HCl — Subjects will be given a single oral dose in tablet form containing 850 mg of metformin
  Other Names: GLUCOPHAGE

SUMMARY:
Specific Aims: To compare metformin pharmacokinetics in monozygotic and dizygotic twin pairs. Comparing renal clearance of metformin in monozygotic and dizygotic twins will allow us to better understand the influence of heredity on variation in renal elimination. Furthermore, genotyping renal transporter genes in monozygotic and dizygotic twin pairs with significant differences in renal clearance of metformin may give us insight into the genes responsible for this variability.

DETAILED DESCRIPTION:
Twin studies have long been a valuable tool for examining the relative role of environment and heredity in health issues such as disease and drug response. For example, twin studies in the 1960's and 1970's showed for the first time that variability in the elimination of many drugs was largely influenced by heredity. Monozygotic twin pairs showed little variability in the elimination of various drugs while dizygotic twin pairs, sharing only about one half of their genes, showed much greater variability. It is now known that the some of the variability in drug elimination observed in dizygotic twins was due to genetic differences in drug metabolizing enzymes, such as the cytochrome P450's. However, genetic variation in other genes, such as membrane transporters may also contribute to variability in drug response.

Membrane transporters play multiple roles in the body; they help to maintain cellular homeostasis through import and export mechanisms and also play an important role in drug response, affecting both the pharmacokinetics and pharmacodynamics of drugs. Animal studies using mice genetically deficient in drug transporters and reports of drug interaction studies involving transporter substrates have provided convincing evidence that the level of function of several important drug transporters is an important determinant of drug response.

The current study will examine differences in the renal clearance of metformin in monozygotic and dizygotic twin pairs. Metformin is an antidiabetic drug that has no significant hepatic metabolism and is actively secreted by the kidneys. Studies in our lab have shown that metformin is a substrate of the human organic cation transporter, hOCT2, which appears to be a major transporter involved in the renal secretion of cationic drugs. Data in the literature indicate that there is substantial variation in the net secretory clearance of metformin in normal, healthy volunteers. In five healthy volunteers, the ratio of renal clearance to creatinine clearance ranged from 1.5 to 4.2, nearly a 3-fold variation. We hypothesize that genetic variation in secretory transporters in the kidney, like hOCT2, may be responsible for the inter-individual differences in the secretory clearance of metformin and other drugs. Studies examining renal clearance of metformin in monozygotic and dizygotic twins will allow us to better understand the influence of heredity on variation in renal elimination. Furthermore, genotyping monozygotic and dizygotic twin pairs with significant differences in renal clearance of metformin may give us insight into the genes responsible for this variability.

ELIGIBILITY:
Inclusion Criteria:

* Part of either a monozygotic or dizygotic twin pair.
* Healthy (by medical history and laboratory values).
* Between 18 and 40 years old.

Exclusion Criteria:

* Taking regular medication other than vitamins.
* Individuals with anemia (hemoglobin < 12 g/dL), an elevation in liver enzymes to higher than double the respective normal value, or elevated creatinine concentrations (males ≥ 1.5 mg/dL, females ≥ 1.4 mg/dL Pregnant at time of study.
* Diagnosis of hypoglycemia, phlebitis and/or stroke will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2001-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To compare metformin pharmacokinetics in monozygotic and dizygotic twin pairs. | 24 hours
  Comparing renal clearance of metformin in monozygotic and dizygotic twins will allow us to better understand the influence of heredity on variation in renal elimination. Furthermore, genotyping renal transporter genes in monozygotic and dizygotic twin pairs with significant differences in renal clearance of metformin may give us insight into the genes responsible for this variability.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Giacomini, PhD, Principal Investigator — University of California San Francsico
Locations (1):
- University of California San Francsico, San Francisco, California, United States

REFERENCES:
- [Background] Leabman MK, Giacomini KM. Estimating the contribution of genes and environment to variation in renal drug clearance. Pharmacogenetics. 2003 Sep;13(9):581-4. doi: 10.1097/00008571-200309000-00007. PMID 12972957
- [Result] Leabman MK, Huang CC, Stryke D, Johns SJ, Kawamoto M, Ferrin TE, DeYoung J, Taylor TR, De La Cruz M, Herskowitz I, Giacomini KM. PharmGKB update: I. Genetic variants of the organic cation transporter 2 (OCT2, SLC22A2). Pharmacol Rev. 2003 Sep;55(3):399. doi: 10.1124/pr.55.3.6. Epub 2003 Jul 17. No abstract available. PMID 12869664